CLINICAL TRIAL: NCT01098786
Title: Observational Study to Evaluate Safety of Cell-derived A/H1N1 Influenza HA Vaccine in Healthy Japanese Subjects
Brief Title: Drug Use Investigation for Cell-culture Derived Influenza A (H1N1) Emulsion HA Vaccine
Status: Completed | Type: Observational
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: V110_11
Record Dates: First submitted 2010-03-31; First posted 2010-04-05 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Swine-Origin Influenza A H1N1 Virus
Keywords: Influenza A; H1N1 subtype; Vaccine; Adjuvant; Cell culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Healthy
  Interventions: Biological: Cell-derived A/H1N1 influenza HA vaccine

INTERVENTIONS:
Biological: Cell-derived A/H1N1 influenza HA vaccine — Single group vaccinated

SUMMARY:
This is to evaluate safety of cell-derived A/H1N1 influenza HA vaccine in healthy Japanese subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy Japanese

Exclusion Criteria:

1. The person has received any other company's new influenza vaccine (swine-derived A/H1N1) before vaccination with this product.
2. The person has participated in any clinical study of this product or any other company's new influenza vaccine (swine-derived A/H1N1) and received the investigational vaccine.

   The person is regarded as a subject in one of the following items 3) to 6) who is not appropriate to receive preventive vaccination as described in the current package insert.
3. The person shows obvious fever.
4. The person obviously suffers from serious acute disease.
5. The person has obviously shown anaphylaxis due to an ingredient of this vaccine.
6. The person is otherwise in an inappropriate state to receive preventive vaccination.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Community sample
Sampling Method: Non-Probability Sample
Enrollment: 556 (Actual)
Dates: Start 2010-02; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Evaluate clinical symptoms according to the subject background after vaccination | 28 days

SECONDARY OUTCOMES:
The kinds, degrees, durations and onset ratios of adverse events | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- National Hospital Organization Kumamoto Medical Center, Chuo-ku, Kumamoto, Japan